CLINICAL TRIAL: NCT01763411
Title: Visual Performance of Pseudophakic Patient With Different Intraocular Lenses
Acronym: ETDRS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Wilson Takashi Hida, MD PhD, Hospital Oftalmologico de Brasilia
Other Study IDs: HOB-12/12; HOB03012013 (Other: Hospital Oftalmologico de Brasilia)
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Cataract; Lens Diseases; Eye Diseases
Keywords: Cataract; Vision; Intraocular lens; Multifocal; Monofocal
MeSH Terms: conditions — Cataract; Lens Diseases; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Multifocal Spheric Intraocular Lens (Restor SN60D3 IOL): No Intervention: Multifocal Spheric IOL implantation
- Monofocal Spheric Intraocular Lens (AcrySof SN60AT IOL): No Intervention: Monofocal Spheric IOL implantation
- Multifocal Aspheric Intraocular Lens (Tecnis ZMA00 IOL): No intervention Multifocal IOL implantation
- Monofocal Aspheric Intraocular Lens (AcrySof SN60WF IOL): No Intervention: Monofocal IOL implantation
- Multifocal Aspheric Intraocular Lens (Tecnis ZMB00 IOL): No intervention Multifocal IOL implantation
- Multifocal Spheric Intraocular Lens (Restor SN6AD1 IOL): No intervention Multifocal IOL implantation

SUMMARY:
This retrospective study comprised patients with cataract, corneal astigmatism, and motivation for spectacle independence. In all cases, a multifocal and monofocal Intraocular Lens was been implanted in the capsular bag. Three months postoperatively, distance, intermediate, and near visual acuities; spherical equivalent; residual refractive astigmatism; defocus curve; and contrast sensitivity was evaluated. A patient-satisfaction and visual phenomena questionnaire was also been administered.

DETAILED DESCRIPTION:
Postoperative evaluation was performed at 3 months. The uncorrected and corrected distance visual acuity were assessed using the 100% contrast Early Treatment Diabetic Retinopathy Study chart, uncorrected intermediate visual acuity at 70 cm, and uncorrected near visual acuity at 40 cm; a binocular defocus curve was constructed using the ETDRS chart at 4 m and adding to the patient's manifest refraction +2.50 to -5.00 D sphere in 0.50 increments. The cylinder axis of the Intraocular lens (IOL) was measured at the slitlamp using the beam protractor after full mydriasis. The mean of the absolute values of degrees the intraocular lens was off axis was determined.

Contrast sensitivity was measured using the CSV-1000 HGT instrument (VectorVision, Inc.), which presents a translucent chart divided into 4 cycles with spatial frequencies of 3, 6, 12 and 18 cycles per degree. The background illumination of the translucent chart does not depend on room lighting. All measurements were obtained under mesopic (5 cd/m2) and photopic (85 cd/m2) conditions. The examinations were performed unilaterally at a distance of 2.5 m with Best-corrected visual acuity (BCVA) and an undilated pupil. All measurements were performed under the same conditions.

Patient satisfaction and quality of life were assessed by a simple questionnaire. Patients were interviewed 3 months postoperative. Patients were asked about visual disturbances, visual lifestyle activities, spectacle use, and satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

Cataract Any race Either gender Diagnosis of cataracts both eyes Pre-existing physical conditions that could skew visual results, such as Diabetes, Retinal detachment, Macular degeneration, or Cancer Subjects must have > 1.00 diopter of astigmatism

Exclusion Criteria:

Central endothelial cell count less than 2000 cells/mm2 glaucoma or intraocular pressure greater than 21 mmHg amblyopia Retinal abnormalities Diabetes mellitus steroid or immunosuppressive treatment Connective tissue diseases

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was derived from patients who had phacoemulsification with multifocal or mono focal intraocular lens (IOL) in Sao Paulo University School of Medicine, Brazil. Patients with senile cataract with vision-impairing disease characterized by gradual, progressive opacity of the lens.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual Performance in Pseudophakic Patients With Different Intraocular Lens | 6 months postoperative
  Postoperative evaluation was been performed at 6 months. The uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) was assessed using the 100% contrast ETDRS chart; a binocular defocus curve was constructed using the ETDRS chart at 4 m.

SECONDARY OUTCOMES:
Contrast sensitivity | 6 months
  Contrast sensitivity was measured using the CSV-1000 HGT instrument (VectorVision, Inc.), which presents a translucent chart divided into 4 cycles with spatial frequencies of 3, 6, 12 and 18 cycles per degree (cpd). The background illumination of the translucent chart does not depend on room lighting. All measurements was obtained under mesopic (5 cd/m2) and photopic (85 cd/m2) conditions. The examinations was performed unilaterally at a distance of 2.5 m with BCVA and an undilated pupil. All measurements was performed under the same conditions.
Patient satisfaction | 6 months
  Patient satisfaction and quality of life was assessed by a simple questionnaire. Patients was interviewed 6 months postoperative. Patients was asked about visual disturbances, visual lifestyle activities, spectacle use, and satisfaction with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson T Hida, MD, Principal Investigator — University of Sao Paulo, Brazil; Newton J Kara-Junior, MD PhD, Study Chair — University of Sao Paulo, Brazil; Celso T Nakano, MD, Principal Investigator — University of Sao Paulo, Brazil; Patrick Tzelikis, MD PhD, Study Director — Hospital Oftalmologico de Brasilia; Mario Augusto D Chaves, MD, Principal Investigator — Hospital Oftalmologico de Brasilia
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Kohnen T, Nuijts R, Levy P, Haefliger E, Alfonso JF. Visual function after bilateral implantation of apodized diffractive aspheric multifocal intraocular lenses with a +3.0 D addition. J Cataract Refract Surg. 2009 Dec;35(12):2062-9. doi: 10.1016/j.jcrs.2009.08.013. PMID 19969209
- [Background] Alfonso JF, Fernandez-Vega L, Orti S, Ferrer-Blasco T, Montes-Mico R. Refractive and visual results after implantation of the AcrySof ReSTOR IOL in high and low hyperopic eyes. Eur J Ophthalmol. 2009 Sep-Oct;19(5):748-53. doi: 10.1177/112067210901900511. PMID 19787593
- [Result] Hida WT, Motta AF, Kara-Jose Junior N, Costa H, Tokunaga C, Cordeiro LN, Gemperli D, Nakano CT. [Comparison between OPD-Scan results and visual outcomes of Tecnis ZM900 and Restor SN60D3 diffractive multifocal intraocular lenses]. Arq Bras Oftalmol. 2008 Nov-Dec;71(6):788-92. doi: 10.1590/s0004-27492008000600004. Portuguese. PMID 19169507
- [Derived] Chaves MA, Hida WT, Tzeliks PF, Goncalves MR, Nogueira Fde B, Nakano CT, Motta AF, Araujo AG, Alves MR. Comparative study on optical performance and visual outcomes between two diffractive multifocal lenses: AMO Tecnis (R) ZMB00 and AcrySof (R) IQ ReSTOR (R) Multifocal IOL SN6AD1. Arq Bras Oftalmol. 2016 May-Jun;79(3):171-6. doi: 10.5935/0004-2749.20160050. PMID 27463628